CLINICAL TRIAL: NCT00084383
Title: A Safety and Efficacy Trial of Lethally Irradiated Allogeneic Pancreatic Tumor Cells Transfected With the GM-CSF Gene in Combination With Adjuvant Chemoradiotherapy for the Treatment of Adenocarcinoma of the Pancreas
Brief Title: Vaccine Therapy Combined With Adjuvant Chemoradiotherapy in Treating Patients With Resected Stage I or Stage II Adenocarcinoma (Cancer) of the Pancreas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J9988; R01CA088058 (NIH); P30CA006973 (NIH); JHOC-J9988
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Results first posted 2013-07-15 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: Pancreatic Cancer
Keywords: stage I pancreatic cancer; stage II pancreatic cancer; duct cell adenocarcinoma of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GVAX pancreatic cancer vaccine (Experimental): 5E8 vaccine cells. The first vaccination is administered 6-8 weeks after surgery. Four to eight weeks following the completion of the last cycle of adjuvant radiation and chemotherapy (chemo-radiation therapy is standard of care and not part of the protocol) eligible patients will receive three additional vaccinations at one month intervals. Patients who continue to remain disease-free will receive a fifth "booster" vaccination, six months following the fourth vaccination
  Interventions: Biological: GVAX pancreatic cancer vaccine

INTERVENTIONS:
Biological: GVAX pancreatic cancer vaccine — Patients will receive vaccinations consisting of 5E8 vaccine cells. The first vaccination is administered 6-8 weeks after surgery. Four to eight weeks following the completion of the last cycle of adjuvant radiation and chemotherapy (chemo-radiation therapy is standard of care and not part of the protocol) eligible patients will receive three additional vaccinations at one month intervals. Patients who continue to remain disease-free will receive a fifth "booster" vaccination, six months following the fourth vaccination.

SUMMARY:
RATIONALE: Vaccines made from gene-modified pancreatic cancer cells may make the body build an immune response to kill tumor cells. Drugs used in chemotherapy, such as fluorouracil, work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Giving vaccine therapy together with chemotherapy and radiation therapy after surgery may kill any remaining tumor cells.

PURPOSE: This phase II trial is studying how well giving vaccine therapy together with adjuvant chemoradiotherapy works in treating patients with resected stage I or stage II adenocarcinoma (cancer) of the pancreas.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine overall and disease-free survival of patients with resected stage I or II adenocarcinoma of the pancreas treated with adjuvant chemoradiotherapy in combination with GVAX pancreatic cancer vaccine.

Secondary

* Correlate specific in vivo parameters of immune response (post-vaccination delayed-type hypersensitivity reactions to autologous tumor, mesothelin-specific T-cell response, and the degree of local eosinophil, macrophage, and T-cell infiltration at the vaccine site) with clinical responses in patients treated with this regimen.
* Determine the toxic effects associated with intradermal injections of this vaccine in these patients.

OUTLINE: This is an open-label study.

* Post surgery vaccination: Within 8-10 weeks after pancreaticoduodenectomy, patients receive GVAX pancreatic cancer vaccine intradermally (ID) on day 0.
* Adjuvant chemoradiotherapy: Within 16-28 days after the first vaccination, patients receive fluorouracil (5-FU) IV continuously for 3 weeks. Approximately 1-2 weeks after completion of 5-FU, patients receive chemoradiotherapy comprising radiotherapy daily and 5-FU IV continuously for 26-28 weeks. Approximately 3-5 weeks after completion of chemoradiotherapy, patients receive 5-FU IV continuously for 4 weeks. 5-FU repeats every 6 weeks for 2 courses.
* Post chemoradiotherapy vaccination: Within 4-8 weeks after the completion of chemoradiotherapy, patients receive GVAX pancreatic cancer vaccine ID on days 0, 28, 56, and 196.

Treatment continues in the absence of unacceptable toxicity.

Patients are followed every 3 months for 1 year and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive ductal adenocarcinoma of the head, neck, and uncinate process of the pancreas

  * Mixed adenocarcinoma tumors allowed if the predominant invasive component of the tumor is adenocarcinoma
  * Stage I or II (clinical stage T1-3, N0-1, M0) disease
* Has undergone pancreaticoduodenectomy at the Johns Hopkins Hospital within the past 8-10 weeks

  * Completely resected (R0) or microscopic residual (R1) disease
* No diagnosis other than ductal adenocarcinoma, including any of the following:

  * Adenosquamous
  * Squamous cell
  * Colloid
  * Islet cell
  * Non-invasive intraductal papillary mucinous neoplasms
  * Serous or mucinous cystadenoma or cystadenocarcinoma
  * Carcinoid
  * Small or large cell carcinoma
  * Intraductal oncocytic papillary neoplasms
  * Osteoclast-like giant cell tumors
  * Acinar cell carcinoma
  * Pancreatoblastoma
  * Solid pseudopapillary tumors
  * Undifferentiated small cell carcinoma
  * Non-epithelial tumors (sarcoma, gastrointestinal stromal tumor, or lymphoma)
  * Adenocarcinoma of the ampulla
  * Adenocarcinoma of the distal bile duct
  * Adenocarcinoma of the duodenum
* No recurrent disease
* No metastatic disease, including peritoneal implants or liver and/or lung involvement

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count >/= 1,500/mm^3
* Platelet count >/= 100,000/mm^3
* Hemoglobin >/= 10 g/dL

Hepatic

* Bilirubin </= 2 mg/dL
* AST/ALT </= 2 times upper limit of normal (ULN)
* Alkaline phosphatase </= 5 times ULN

Renal

* Creatinine </= 2 mg/dL

Pulmonary

* No asthma or chronic obstructive pulmonary disease requiring systemic corticosteroids

Immunologic

* HIV negative
* No active infection
* No prior or concurrent autoimmune disease requiring treatment with systemic immunosuppressants, including any of the following:

  * Inflammatory bowel disease
  * Systemic vasculitis
  * Scleroderma
  * Psoriasis
  * Multiple sclerosis
  * Hemolytic anemia or immune thrombocytopenia
  * Rheumatoid arthritis
  * Systemic lupus erythematosus
  * Sjogren's syndrome
  * Sarcoidosis
* Negative results to viral delayed-type hypersensitivity serology testing if autologous tumor cells are available

Other

* No postoperative complications (e.g., inability to take oral nutrition >/= 1,500 calories/day, ongoing requirement for long-term biliary stenting, or persistence of wound infection)
* No other malignancy within the past 5 years except nonmelanoma skin cancer
* No uncontrolled medical conditions that would preclude study participation
* No other major active medical or psychosocial problem that could be exacerbated by study treatment
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 4 weeks after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 1 month since prior biologic therapy
* No other concurrent biologic therapy, immunotherapy, or gene therapy for pancreatic cancer

Chemotherapy

* More than 1 month since prior chemotherapy
* No other concurrent chemotherapy for pancreatic cancer

Endocrine therapy

* More than 28 days since prior systemic steroids
* No concurrent systemic corticosteroids

Radiotherapy

* More than 1 month since prior radiotherapy
* No other concurrent radiotherapy for pancreatic cancer

Surgery

* See Disease Characteristics
* Recovered from prior surgery

Other

* More than 1 month since prior participation in an investigational new drug trial
* No other concurrent investigational therapy for pancreatic cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2002-01; Primary Completion 2005-12 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A. Laheru, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Lutz E, Yeo CJ, Lillemoe KD, Biedrzycki B, Kobrin B, Herman J, Sugar E, Piantadosi S, Cameron JL, Solt S, Onners B, Tartakovsky I, Choi M, Sharma R, Illei PB, Hruban RH, Abrams RA, Le D, Jaffee E, Laheru D. A lethally irradiated allogeneic granulocyte-macrophage colony stimulating factor-secreting tumor vaccine for pancreatic adenocarcinoma. A Phase II trial of safety, efficacy, and immune activation. Ann Surg. 2011 Feb;253(2):328-35. doi: 10.1097/SLA.0b013e3181fd271c. PMID 21217520

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GVAX Pancreatic Cancer Vaccine
Started | 60
Completed | 13
Not Completed | 47

BASELINE CHARACTERISTICS:
Arm/Group | GVAX Pancreatic Cancer Vaccine
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 27
Age Continuous [Mean (Standard Deviation); unit: years] | 62 (9.375)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 37
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival in patients treated with adjuvant chemoradiotherapy in sequence with the irradiated allogeneic GM-CSF transfected pancreatic tumor cell lines. Overall survival is defined as time from surgery until death, regardless of cause.
Time Frame: Participants were followed for the duration of the study, an average of 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | GVAX Pancreatic Cancer Vaccine
Number analyzed (Participants) | 60
Months | 24.8 [21.2 to 31.6]

2. Secondary Outcome: To Further Identify and Characterize Toxicities Associated With Intradermal Injections of the Vaccine That Were Initially Reported in the Phase 1 Trial.
Time Frame: 4 years
Reporting Status: Not Posted

3. Secondary Outcome: Estimate the Association of Specific in Vivo Parameters of Immune Response With Clinical Responses in Patients Treated With Combination Chemoradiotherapy Together With the Irradiated Allogeneic GM-CSF Transfected Pancreatic Tumor Cell Lines.
Description: The specific immune parameters include: post-vaccination delayed type hypersensitivity reactions to autologous tumor and the degree of local eosinophil, macrophage, and T cell infiltration at the vaccine site, and mesothelin-specific T cell responses.
Time Frame: Continuous
Reporting Status: Not Posted

4. Primary Outcome: Disease-free Survival
Description: Disease-free Survival in Patients Treated With Adjuvant Chemoradiotherapy in Sequence With the Irradiated Allogeneic GM-CSF Transfected Pancreatic Tumor Cell Lines. DFS is defined as time from surgery until clinical evidence of disease (eg, CT scan) or death due to any cause.
Time Frame: Participants were followed for the duration of the study, an average of 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | GVAX Pancreatic Cancer Vaccine
Number analyzed (Participants) | 60
Months | 17.3 [14.6 to 22.8]

ADVERSE EVENTS:
Arm/Group | GVAX Pancreatic Cancer Vaccine
Serious Adverse Events (participants affected / at risk) | 2/60
Other Adverse Events (participants affected / at risk) | 60/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | GVAX Pancreatic Cancer Vaccine (N=60)
Pain, Cancer related (Hepatobiliary disorders) | 1/1 (1)
Biliary Obstruction, secondary to progessive disease (Hepatobiliary disorders) | 1/1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GVAX Pancreatic Cancer Vaccine (N=60)
Eosinophils, elevated (Blood and lymphatic system disorders) | 17 (30)
Chills (General disorders) | 11 (12)
Fatigue (General disorders) | 9 (11)
Fever (General disorders) | 11 (19)
Flu like symptoms (General disorders) | 7 (13)
Blister (Skin and subcutaneous tissue disorders) | 4 (4) — Localized vaccine site reaction
Erythema (Skin and subcutaneous tissue disorders) | 60 (172) — Localized vaccine site reaction
Induration (Skin and subcutaneous tissue disorders) | 60 (171) — Localized vaccine site reaction
Pruritis (Skin and subcutaneous tissue disorders) | 51 (152) — Localized vaccine site reaction
Tenderness (Skin and subcutaneous tissue disorders) | 55 (142) — Localized vaccine site reaction
Vaccine site flare (Skin and subcutaneous tissue disorders) | 7 (12) — Localized vaccine site reaction
Rash (Skin and subcutaneous tissue disorders) | 7 (13)
Nausea (Gastrointestinal disorders) | 7 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (12)
Dizziness (Nervous system disorders) | 3 (4)
Headache (Nervous system disorders) | 5 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes